CLINICAL TRIAL: NCT02277366
Title: A Multi-center Randomized Control Study of Bronchoscopy in Early Lung Cancer Screening of High Risk Population
Brief Title: Role of Bronchoscopy in Early Lung Cancer Screening of High Risk Population
Status: Terminated | Type: Observational
Why Stopped: We have recruited some patients, but we haven't found any significant result by bronchoscopy in the high risk population.
Sponsor: Tang-Du Hospital (Other)
Collaborators: Changhai Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Xinqiao Hospital of Chongqing (Other); China Meitan General Hospital (Other); Micro-Tech (Nanjing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: lungcancer screening; 201402024-BS (Other Grant/Funding Number: Ministry of Health in China)
Record Dates: First submitted 2014-10-21; First posted 2014-10-29 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Lung Neoplasms
Keywords: Lung Neoplasms; Bronchoscopy; Early Detection of Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Fluorescence/Narrow Band Bronchoscopy: All patients in the group are examined by Fluorescence Bronchoscopy and Narrow Band Bronchoscopy to make a early detection of lung cancer.
  Interventions: Procedure: Fluorescence Bronchoscopy/Narrow Band Bronchoscopy
- Routine Bronchoscopy: All patients in this group are examined by routine bronchoscopy to make a early detection of lung cancer.

INTERVENTIONS:
Procedure: Fluorescence Bronchoscopy/Narrow Band Bronchoscopy — Fluorescence Bronchoscopy and Narrow Band Bronchoscopy are used in the Fluorescence/Narrow Band Bronchoscopy group to make a diagnosis of lung cancer.
  Groups: Fluorescence/Narrow Band Bronchoscopy

SUMMARY:
The purpose of this study is to determine the diagnostic yield of early lung cancer in high risk population, who smokes or has other risk factors, by different bronchoscopy,. Furthermore, another purpose is to determine whether the different bronchoscopy are significant different in diagnosing early lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient is over 40 years in age and is a heavy cigarette smoker.(smoking index is over 400)
* Patient has been coughing irritably for 2-3 weeks with a failed treatment and without obvious causes.
* The nature of cough changes in a patient who has chronic respiratory disease.
* Patient has blood-stained sputum persistently or repeatedly without obvious causes.

Patient will be included if accorded with any item of above.

Exclusion Criteria:

* Patient has dysrhythmia or cardiovascular disease that poses a risk during exercise.
* Patient has uncontrollable hypertension (SBP > 180mmHg).
* Patient has severe organ dysfunction (shock, severe hepatic and renal dysfunction, massive hemorrhage of upper gastrointestine, diffuse intravascular coagulation(DIC) and massive hemoptysis,etc).
* Patient has blood coagulation disorders (PT>2 times the upper limit of normal(ULN) or Platelet(PLT)<50000/ul）.
* Patient has severe dyspnea.
* Patient is allergic to local anesthetic.
* Patient is unable to provide informed consent.
* Patient is not an appropriate candidate for or is unable to tolerate flexible bronchoscopy procedures.
* Patient has any disease or condition that interferes with completion of initial or follow-up assessments of the effectiveness endpoints.
* Patient has demonstrated unwillingness or inability to complete screening or baseline data collection procedures.
* Patient participated in a study of an investigational drug or device within the past 30 days prior to participation in this study, or is currently participating in another clinical study.
* Patient has pulmonary lesions suspected to be cancer from CT images.
* Female patient of childbearing potential has a positive result from a pregnancy test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients recruited in the study should meet one item as follows.
  * Patient is over 40 years in age and is a heavy cigarette smoker.(smoking index is over 400.)
  * Patient has been coughing irritably for 2-3 weeks with a failed treatment and without obvious causes.
  * The nature of cough changes in a patient who has chronic respiratory disease.
  * Patient has blood-stained sputum persistently or repeatedly without obvious causes.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-05; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of Lung Cancer | 1 week

SECONDARY OUTCOMES:
Number of Participants with Serious Adverse Events | 1 week

OTHER OUTCOMES:
Cost of all examinations to make a diagnosis | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Faguang Jin, Ph.D, MD, Principal Investigator — Tang-Du Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Moghissi K, Dixon K, Stringer MR. Current indications and future perspective of fluorescence bronchoscopy: a review study. Photodiagnosis Photodyn Ther. 2008 Dec;5(4):238-46. doi: 10.1016/j.pdpdt.2009.01.008. Epub 2009 Feb 23. PMID 19356663
- [Background] Ali AH, Takizawa H, Kondo K, Nakagawa Y, Toba H, Khasag N, Kenzaki K, Sakiyama S, Mohammadien HA, Mokhtar EA, Tangoku A. Follow-up using fluorescence bronchoscopy for the patients with photodynamic therapy treated early lung cancer. J Med Invest. 2011 Feb;58(1-2):46-55. doi: 10.2152/jmi.58.46. PMID 21372486
- [Background] Edell E, Lam S, Pass H, Miller YE, Sutedja T, Kennedy T, Loewen G, Keith RL, Gazdar A. Detection and localization of intraepithelial neoplasia and invasive carcinoma using fluorescence-reflectance bronchoscopy: an international, multicenter clinical trial. J Thorac Oncol. 2009 Jan;4(1):49-54. doi: 10.1097/JTO.0b013e3181914506. PMID 19096306
- [Background] Venmans BJ, Van Boxem TJ, Smit EF, Postmus PE, Sutedja TG. Results of two years expenience with fluorescence bronchoscopy in detection of preinvasive bronchial neoplasia. Diagn Ther Endosc. 1999;5(2):77-84. doi: 10.1155/DTE.5.77. PMID 18493485
- [Background] Gabrecht T, Lovisa B, van den Bergh H, Wagnieres G. Autofluorescence bronchoscopy: quantification of inter-patient variations of fluorescence intensity. Lasers Med Sci. 2009 Jan;24(1):45-51. doi: 10.1007/s10103-007-0518-y. Epub 2007 Nov 30. PMID 18060444